CLINICAL TRIAL: NCT07041918
Title: Evaluation of the Performance and Safety of VACUSERA® PRP Tubes in the Preparation of Autologous Platelet-Rich Plasma: A Prospective, Observational Medical Device Study (PMCF)
Brief Title: Evaluation of the Performance and Safety of VACUSERA® PRP Tubes in the Preparation of Autologous Platelet-Rich Plasma
Acronym: PRP
Status: Completed | Type: Observational
Sponsor: Disera Tıbbi Cihazlar Lojistik Sanayi ve Ticaret A.Ş (Industry)
Responsible Party: Sponsor
Other Study IDs: 0.PRT.KGV.002
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: No Disease or Condition is Being Studied

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: The study is entirely designed to analyze product performance (analyze only results from whole blood and derived from the PRP tubes), and no interventions will be performed. — The study will evaluate and analyze only the results obtained from whole blood in the hemogram test and the results derived from the PRP tubes. The main objective is to measure the performance of the Vacusera PRP Tube and Vacusera PRP Tube with Gel in obtaining platelet-rich plasma. The study is entirely designed to analyze product performance, and no interventions will be performed.

SUMMARY:
Study Design After the eligibility assessment during screening and obtaining a written informed consent form, the volunteers' demographic information and medical history will be recorded.

In addition to the hemogram and pregnancy test to be performed on the volunteers in this study, an additional tube (approximately 8 ml (±10%) for the VACUSERA® Single PRP Tube or approximately 7 ml (±10%) for the VACUSERA® Single Gel PRP Tube) will be used to obtain platelet-rich plasma (PRP). After centrifugation of the PRP tubes, the platelet (PLT) count in the resulting plasma will be analyzed, and the concentration increase in relation to whole blood will be evaluated.

DETAILED DESCRIPTION:
The study is a post-market clinical follow-up (PMCF) study aimed at proving the effectiveness and safety of PRP tubes that are already CE (European Conformity) certified and released on the market. After the eligibility assessment during screening and obtaining the written informed consent form, the demographic information and medical history of eligible volunteers will be recorded on a paper case report form.

The analysis conducted using the G-Power power test calculated that the number of patients to be included in the study is 194.In addition to the hemogram and pregnancy test to be performed on the volunteers in this study, an additional tube (approximately 8 ml (±10%) for the VACUSERA® Single PRP Tube or approximately 7 ml (±10%) for the VACUSERA® Single Gel PRP Tube) will be used to obtain platelet-rich plasma (PRP). After centrifugation of the PRP tubes, platelet (PLT) count will be performed on the obtained plasma, and the concentration increase relative to whole blood will be analyzed.

Screening Day (Day 1):

Volunteers will undergo a medical history review to check eligibility for inclusion in the study.

Analysis Day (Day 1):

A single blood sample will be collected for platelet (hemogram) testing, and for women of reproductive age, a beta HCG (human chorionic gonadotropin) test will be conducted.

Platelet (PLT) count will be performed on the plasma obtained from the blood sample collected in the PRP tubes.

The concentration increase in the resulting plasma will be analyzed in relation to whole blood.The PRP results of volunteers who do not meet the inclusion criteria based on hemogram test results or who are pregnant will not be included in the study.

ELIGIBILITY:
INCLUSION CRITERIA

Male or female volunteers between the ages of 18 and 60, as defined in the target population during screening,

Body Mass Index (BMI) between 18 and 32 during screening,

No pregnancy or risk of pregnancy for women,

Willing to participate and provide written informed consent and comply with the study restrictions,

Must not have participated in any clinical trial within 2 months prior to the start of the study,

Must be able to communicate with the researcher or authorized personnel.

EXCLUSION CRITERIA

Platelet dysfunction syndrome,

Critical thrombocytopenia,

Hemodynamic instability,

Septicemia,

Local infection at the site of the procedure,

Autoimmune diseases,

History of chronic infections,

Chronic liver pathology,

Patients receiving anticoagulant/antiplatelet therapy,

Use of NSAIDs (except for paracetamol) in the last 7-10 days,

History of alcohol and/or drug addiction,

Corticosteroid use,

Fever or illness in the past week,

Cancer (especially blood and bone cancers),

Hemoglobin (HGB) levels below 10 g/dl or above 16.5 g/dl in men and 16 g/dl in women,

Platelet count below 105/μl,

Those under immunosuppressive therapy,

Any condition or disease detected during the medical interview/physical examination that, in the opinion of the researcher or designated personnel, would make the volunteer unsuitable for the study, put them at unnecessary risk, or interfere with the volunteer's ability to complete the study,

Clinically significant deviation from normal findings in the physical examination, including vital signs,

Patients planning pregnancy or not using contraception,

Patients using hormonal contraceptive methods to prevent pregnancy,

Breastfeeding women,

Poor venous access for blood sampling,

Plasma or blood donation within the last 2 months,

It is recommended to select patients who do not use tobacco products during the study, as it is considered that it may affect the product's performance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male or female volunteers between the ages of 18 and 60, as defined in the target population during screening,
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Increasing platelet concentration | Day 1: Blood will be taken on the same day and sent for analysis for counting.
  Approximately 8 ml (±10%) of blood will be collected to the PRP Tubes and approximately 7 ml (±10%) to the PRP Tube with Gel, and platelet (PLT) count will be performed on the obtained plasma, with the concentration increase relative to whole blood analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Recep Selim Şentürk, MD, Principal Investigator — Medical Point Hastanesi Klinik Araştırmalar Merkezi
Locations (1):
- Medical Point Hastanesi Klinik Araştırmalar Merkezi, Izmir, Karşıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No